CLINICAL TRIAL: NCT00111202
Title: Schizophrenia and Genetic Counseling: A Survey of People With Schizophrenia and Their Relatives
Brief Title: Schizophrenia and Genetic Counseling
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sarah Lawrence College (Other)
Other Study IDs: SLC1012005
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2005-09-30 (Estimated); Status verified 2005-05

CONDITIONS: Schizophrenia
Keywords: Genetic counseling; Genetic counselling; Genetics; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This research is designed to investigate the perceptions and opinions of individuals who either have schizophrenia or who have a family member with schizophrenia, in relation to genetic counseling. Data will be collected via a 15 minute online questionnaire. There is also an option for respondents to participate in a 45 minute interview if they wish.

It is expected that the study will show that adequate information about genetic counseling is not provided to these individuals. It is also hoped that this research will help to make genetic counseling sessions more specific to people with schizophrenia in their family.

DETAILED DESCRIPTION:
For more information please go to the following website:

http://schizophreniageneticcounseling.blogspot.com

ELIGIBILITY:
Inclusion Criteria:

* anyone diagnosed with schizophrenia OR who has family member diagnosed with schizophrenia
* Over 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-05; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Study Completed, Principal Investigator — SLC